CLINICAL TRIAL: NCT04787887
Title: A Randomized, Double-blind, 2-treatment, 2-period, Crossover Phase I Study to Compare the PK, Safety and Tolerability of 60 IU/kg of Abcertin, and EU-sourced Cerezyme® in Healthy Volunteers Following a Single Intravenous Administration
Brief Title: A Phase I Study to Compare Abcertin and EU-sourced Cerezyme® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISU302-005; ACTRN12619001399189p (Registry Identifier: ANZCTR)
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Gaucher Disease
Keywords: Gaucher Disease; ISU ABXIS Co., Ltd.; ISU302
MeSH Terms: conditions — Gaucher Disease | interventions — Abcertin; imiglucerase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abcertin (Active Comparator): Abcertin 60IU/kg
  Interventions: Drug: Abcertin; Drug: EU-sourced Cerezyme
- Cerezyme (Active Comparator): EU-sourced Cerezyme
  Interventions: Drug: Abcertin; Drug: EU-sourced Cerezyme

INTERVENTIONS:
Drug: Abcertin — 60IU/kg Single Intravenous Administration
  Other Names: Imiglucerase
Drug: EU-sourced Cerezyme — 60IU/kg Single Intravenous Administration
  Other Names: Imiglucerase

SUMMARY:
Primary Objective:

To compare the pharmacokinetics of Abcertin to the reference product, EU-sourced Cerezyme, after single intravenous administration of 60 IU/kg.

Secondary Objective:

To compare the safety, tolerability and immunogenicity of Abcertin to the reference formulation, EU-sourced Cerezyme, after single intravenous administration of 60 IU/kg.

DETAILED DESCRIPTION:
This is a phase 1, single-center, randomized, double-blind, two-way crossover study employing Abcertin and EU-sourced Cerezyme in healthy volunteers between the ages of 18 and 45 years (inclusive). The study aimed to evaluate the PK, safety, tolerability and immunogenicity of Abcertin compared with EU-sourced Cerezyme when administered as a single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have been able to give voluntary written informed consent prior to any study-related procedures.
2. Subject must have been available for the entire study period.
3. Subject was male or female aged between ≥ 18 and ≤ 45 years old.
4. Subject had a body mass index (BMI) between ≥ 18.50 and ≤ 30.00 kg/m2 and weighed between 55 and 105 kg, inclusive.
5. Female subject of childbearing potential must have been non-pregnant and non-lactating and must have had a negative pregnancy test at Screening and at each admission to the clinical research center.
6. Female subject of childbearing potential, with a fertile male sexual partner, must have used adequate contraception from Screening until 90 days after the Follow-up Visit. Adequate contraception is identified as using hormonal contraceptives or an intrauterine device combined with at least one of the following forms of contraception: a diaphragm or cervical cap, or a condom.
7. Male subject must have used adequate contraception and must not have donated sperm from first admission to the clinical research center until 90 days after the Follow-up Visit. Adequate contraception for the male subject and his female partner is defined as using hormonal contraceptives or an intrauterine device combined with at least one of the following forms of contraception: a diaphragm or cervical cap, or a condom.
8. Subject must have been healthy, as determined by the Principal Investigator, based on medical history, physical examination, 12-lead ECG and laboratory evaluations (hematology, blood chemistry, coagulation and urinalysis tests).
9. All values for the subject's clinical laboratory tests of blood and urine should not have been clinically significant, as judged by the Principal Investigator.

Exclusion Criteria:

1. Intake of any investigational drug in another study within 30 days (or 5 half-lives, whichever was greater) prior to the intake of the IP in this study or had received the last dose of IP more than 30 days prior (or 5 half-lives, whichever was greater) but who were on extended follow-up, or planned intake of an investigational drug (other than for this study) during the course of this study.
2. With ongoing symptoms that had indicated acute diseases within 28 days prior to IP administration; acute disease referred to any new onset of symptoms/signs or diagnosis of disease, whether infectious, inflammatory, traumatic, etc., in origin (regardless of whether or not the subject was hospitalized).
3. With any medical history that might have affected IP distribution, metabolism and excretion (e.g., hepatic or renal disease).
4. Positive screen on hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibodies or anti-human immunodeficiency virus (HIV) type 1 and type 2 antibodies. If a potential subject was considered by the Investigator to have false positive result (e.g., HIV antibodies) at Screening, a repeat test should have been done as soon as possible and if the retest was negative, the subject could have been considered eligible for the study.
5. Had clinically significant hypersensitivity or severe allergic reactions (either spontaneous or following IP administration), also including known or suspected clinically relevant drug hypersensitivity to any components of the IP or comparable drugs, including Latex.
6. Had vaccination within 3 months prior to the first IP administration or planned a vaccination before the Follow-up Visit.
7. Safety laboratory tests with the following results:

   1. Aspartate aminotransferase (AST, also known as serum glutamic-oxaloacetic transaminase) or alanine aminotransferase (ALT, also known as serum glutamic-pyruvic transaminase) > 1.5 times the upper limit of normal (ULN), or
   2. Total bilirubin (TBL) > 1.5 times ULN.
8. Subject who had immune deficiency or medication with immunosuppressive agents.
9. Treatment with any medication, prescribed or over-the-counter (OTC) products including herbal remedies, within 14 days prior to Day 1 or longer if the medication had a long half-life, unless agreed as not clinically significant by the Investigator and Sponsor. Exceptions: hormonal contraceptives, acetaminophen ≤ 3 g/day, vitamins at daily recommended doses.
10. Had donated whole blood products (e.g., plasma, platelets) within 60 days, or transfused within 20 days before Screening.
11. History of alcohol or drug abuse or drug addiction (including cannabis products) within the last 12 months before Screening.
12. Subject was willing to comply with the alcohol restrictions. The subject should have refrained from drinking any alcohol within 72 hours prior to Day -1 and should not have consumed more than 3 - 4 units of alcohol per day, to a maximum of 14 units of alcohol per week (1 unit of 10 mL of pure alcohol is equal to 12 ounces [360 mL] of beer, 5 ounces [150 mL] of wine or 1.5 ounces [45 mL] of 80-proof distilled spirits) throughout the study.
13. Heavy smoker (> 5 cigarettes/day) or the subject could not stop smoking during the study period while inpatient at the clinical research center.
14. Positive tests for drugs of abuse or alcohol at Screening or Day -1 (admission to the clinical research center).
15. Family member or employee of the Investigator or clinical research center staff or study team.
16. Those who were not suitable for participation in the study based on the Investigator's judgement, for any reason including laboratory test results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Area under the concentration-time curve (AUC) from time zero to time infinity

SECONDARY OUTCOMES:
Cmax | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Maximum plasma concentration
tmax | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Time to Cmax
AUC0-last | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  AUC from time zero to the time of the last measurable plasma concentration
t½ | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Terminal half-life
CL | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Total body clearance
Vz | Predose(0 minute), during infusion(10, 20, 40, 60, 90, 120 minutes), and after infusion( 5, 10, 20, 30, 40, 50, 60 ,70, 80, 90, 120 minutes)
  Volume of distribution based on the terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, MD, Principal Investigator — Scientia Clinical Research Limited
Locations (1):
- Scientia Clinical Research Limited, Randwick, New South Wales, Australia